CLINICAL TRIAL: NCT01324180
Title: A Phase I Window, Dose Escalating and Safety Trial of Metformin in Combination With Induction Chemotherapy in Relapsed Refractory Acute Lymphoblastic Leukemia: Metformin With Induction Chemotherapy of Vincristine, Dexamethasone, Doxorubicin, and PEG-asparaginase (VPLD)
Brief Title: Vincristine, Dexamethasone, Doxorubicin, and PEG-asparaginase (VPLD) and Metformin for Relapsed Childhood Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pediatric Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16601; Sunshine Project 001 (Other Grant/Funding Number: Pediatric Cancer Foundation)
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; Relapsed; Refractory
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Metformin; Vincristine; Dexamethasone; Calcium Dobesilate; pegaspargase; Polyethylene; Doxorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VLPD Regimen (Experimental): Induction will consist of vincristine, dexamethasone, doxorubicin and PEG asparaginase (so called VPLD - dexamethasone is substituted for prednisone and PEG asparaginase is substituted for L-asparaginase) in combination with metformin. Eligible patients will receive 24 hours of metformin followed by induction. Intrathecal chemotherapy with standard dose cytarabine will be administered at the start of each cycle, with central nervous system (CNS) therapy afterwards determined by findings on staging lumbar puncture.
  Interventions: Drug: Metformin; Drug: Vincristine; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Intrathecal chemotherapy

INTERVENTIONS:
Drug: Metformin — Will be dosed orally BID as per dose level of subject as defined in dose escalation schema. Both liquid and tablet forms are allowed and can be chosen based on convenience. Metformin will be continued throughout the cycle until Day 28 or until the patient is removed from study (e.g. to pursue new lines of therapy such as transplant), whichever occurs sooner.
Drug: Vincristine — 1.5 mg/m^2/dose IV push (maximum single dose 2 mg) on days 2, 9, 16 and 23
  Other Names: Oncovin®; VCR; LCR; NSC #67574
Drug: Dexamethasone — * 10 mg/m^2/day divided BID
  * Take dexamethasone by mouth days 2-15
  Other Names: Decadron®; Hexadrol®; Dexone®; Dexameth®; NSC #34521 (112004)
Drug: PEG-asparaginase — * 2500 IU's/m^2/day
  * Intramuscular injection (IM) or intravenous infusion per institutional standard on days 3, 9, 16 and 23
  * If the patient develops an allergic reaction to PEG while being treated on this protocol, eliminate all future doses of PEG and substitute Erwinia if not intolerant of Erwinia and has no history of pancreatitis.
  * Patients will receive Erwinase® 25,000 IU/m^2 x 6 doses intramuscularly (IM) on a Monday/Wednesday/Friday schedule as a replacement for each scheduled dose of PEG-asparaginase on the original protocol.
  Other Names: Oncaspar; NSC #644954; Pegaspargase; Oncaspar®; Polyethylene; Glycol Conjugated L-asparaginase-H
Drug: Doxorubicin — 60 mg/m^2/day IV over 15 minutes on day 2
  Other Names: Adriamycin®; NSC #123127 (102004)
Drug: Intrathecal chemotherapy — IT cytarabine given intrathecally to all patients on day 1 of each cycle. Dose defined by age. May be given with staging lumbar puncture before enrollment, but must be within 72 hours of starting therapy. If not done at study entry or before, may be done on Day 2 prior to doxorubicin administration.
  * 30 mg for patients age 1-1.99
  * 50 mg for patients age 2-2.99
  * 70 mg for patients greater than 3 years of age IT methotrexate given Intrathecally to all patients who are CNS negative at study entry on day 16 at the dose defined by age.
  Other Names: Cytosine Arabinoside; Ara-C; Cytosar®; NSC #63878 (102004)

SUMMARY:
H. Lee Moffitt Cancer Center and Research Institute will be the Sunshine Project Coordinator, but will not be recruiting locally.

The purpose of the trial is to study the clinical and biological effects of metformin in combination with standard systemic chemotherapy in a disease (relapsed ALL) that has a dismal outcome, as well as to do a dose escalation study to find the Maximum Tolerated Dose (MTD) of metformin in conjunction with ALL therapy. There have also been analysis of patients enrolled on trials who were diabetics on metformin and their outcome was better than patients on the same trial that were not on metformin as their antihyperglycemic.

DETAILED DESCRIPTION:
This will be a phase I protocol of Vincristine, Dexamethasone, Doxorubicin, and PEG-asparaginase (VPLD) and metformin conducted in the Sunshine Project sites for children with recurrent ALL. All sites will be eligible to open this study, provided they agree to adhere to all study procedures and make a good faith effort to obtain all pharmacodynamic and pharmacokinetic evaluations requested.

ELIGIBILITY:
Inclusion Criteria:

* ALL or lymphoblastic lymphoma patients in first or higher relapse.
* Male or Female age 1-30 years at initial diagnosis.
* Signed informed consent.
* Karnofsky / Lansky score above 50%.
* No known contraindications to intended therapies.
* Prior anthracycline exposure: Patients must have had less than 350 mg/m^2 lifetime exposure of anthracycline chemotherapy.
* It must be at least 6 months since the last treatment with a "VPLD" induction/re-induction type regimen (i.e. anthracycline, steroid, asparaginase and vincristine).
* Patients must have adequate organ function.

  * Adequate renal function defined as serum creatinine < 1.5 x upper limit of normal (ULN) for age.
  * Total bilirubin < 1.5 X ULN for age.
  * Alanine transaminase (ALT) < 5 X ULN for age, unless the elevation is disease-related.
  * Adequate cardiac function as defined as shortening fraction of > 27% by echocardiogram or ejection fraction > 45% by gated radionuclide study.

Exclusion Criteria:

* Significant renal impairment as determined per investigator discretion.
* Patients planning on receiving other investigational agents while on this study.
* Patients planning on receiving other anti-cancer therapies while on this study.
* Patients with active infection defined as: positive blood culture within 48 hours of study registration; need for supplemental oxygen or vasopressors within 48 hours of study entry.
* Patient receiving corticosteroids, aside from dexamethasone treatment directed at leukemia.
* Known intolerance to doxorubicin, metformin, or vincristine.
* Patients who have started protocol therapy prior to enrollment. Patient may still enroll if IT therapy was given within 72 hours of study enrollment as part of the diagnostic lumbar procedure.
* Patients may be on hydroxurea until the first dose of metformin is to be given.
* Patients who have a need to continue hydroxurea while on study (Patients may continue on hydroxurea only until the first dose of metformin is to given).
* Patients with creatinine more than 1.5 x the ULN
* Patients must have recovered from the acute side effects of all prior anticancer therapy.

  * At least 1 week from prior cytotoxic chemotherapy.
  * At least 4 weeks from craniospinal irradiation.
  * At least 4 months since hematopoietic stem cell transplant (HSCT) with no evidence of active graft-versus-host disease (GVHD).
* Pregnant or lactating women.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2011-07-18 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 45 days
  MTD determined by Dose Limiting Toxicity (DLT), any time during the first course of therapy. Dose Limiting Toxicities: Any Grade 3 or 4 non-hematological toxicity by Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0 felt to be probably or definitely related to the study agent, persistent marrow aplasia at day 44, lactic acidosis for grade 3 or 4, grade 3 and 4 hypoglycemia.

SECONDARY OUTCOMES:
The Number of Participants with Complete Remission | 45 days
  Patients who have:
  * No evidence of circulating blasts or extramedullary disease;
  * A bone marrow with <5% blasts (M1 marrow); and
  * Recovery of peripheral counts (platelets ≥75,000 and absolute neutrophil count (ANC) ≥750)
    * Qualifying marrow and peripheral counts should be performed within 1 week of each other
The Number of Participants with Biological Response to Treatment | 45 days
  To evaluate the biological response of ALL blasts from children receiving metformin in a window fashion and in later time points.
The Number of Participants with Adverse Events as a Measure of Safety and Feasibility | 45 Days
  To demonstrate the safety and feasibility of the addition of metformin to induction chemotherapy for recurrent ALL.

CONTACTS AND LOCATIONS:
Overall Officials: Julio M. Barredo, M.D., Study Chair — Holtz Children's Hospital University of Miami Miller School of Medicine; Damon Reed, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (5):
- United States (5):
  - Holtz Children's Hospital University of Miami Miller School of Medicine, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Montefiore Medical Center, The Children's Hospital at Montefiore, The Bronx, New York
  - Nationwide Children's Hospital, Columbus, Ohio